CLINICAL TRIAL: NCT03400488
Title: A Phase 1, Randomized, Single-blind, Placebo-controlled Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AZD5718 After Single and Multiple Ascending Dose Administration to Healthy Japanese Men
Brief Title: A Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AZD5718 After Single and Multiple Ascending Dose Administration to Healthy Japanese Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D7550C00004
Record Dates: First submitted 2017-12-12; First posted 2018-01-17 (Actual); Last update posted 2018-06-15 (Actual); Status verified 2018-06

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease,; Cardiovascular disease (CAD),; 5-lipoxygenase activating protein (FLAP) inhibitor,; Leukotrienes.
MeSH Terms: conditions — Coronary Artery Disease; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Masking Description: This study is single-blind (in which the study centre staff will remain blinded during the clinical conduct of a given cohort) with regard to treatment (AZD5718 or placebo) at each dose level. In the event of a medical emergency when management of a subject's condition requires knowledge of the trial medication, the treatment received may be revealed by personnel authorized by the Principal Investigator (PI).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AZD5718 (Experimental): Randomized subjects will receive orally once daily dose of AZD5718 oral suspension on Day 1 (SAD) and MAD from Days 3 to 10. On Day 2, no dose will be given. These procedures will be repeated in all cohorts.
  Interventions: Drug: AZD5718 oral suspension
- Placebo (Placebo Comparator): Randomized subjects will receive orally once daily dose of placebo matching AZD5718 oral suspension on Day 1 (SAD) and MAD form Days 3 to 10. On Day 2, no dose will be given. These procedures will be repeated in all cohorts.
  Interventions: Other: Placebo matching AZD5817 oral suspension

INTERVENTIONS:
Drug: AZD5718 oral suspension — In all cohorts, randomized subjects will receive orally AZD5718 oral suspension SAD (60 mg) on Day 1 and MAD (180 mg, 360 mg and 600 mg) from Days 3 to 10. On Day 2, no dose will be given. In total each subject will receive 9 doses of AZD5718.
  Arms: AZD5718
Other: Placebo matching AZD5817 oral suspension — In all cohorts, randomized subjects will receive orally placebo matching AZD5718 oral suspension on Day 1 and from Days 3 to 10. On Day 2, no dose will be given.
  Arms: Placebo

SUMMARY:
This is a Phase I study to investigate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of the novel compound, AZD5718 in healthy Japanese men. The results from this study will form the basis for decisions on future studies.

DETAILED DESCRIPTION:
This study will be a Phase 1, randomized, single-blind, placebo-controlled, single and multiple ascending dose sequential group design in up to 48 healthy male Japanese subjects, performed at a single study center. The planned number of cohorts is 4 but up to 6 cohorts may be included if the Safety Review Committee (SRC) considers it necessary to repeat a dose level or if additional dose steps are required. Screening will be completed between Days -28 and -1. Primarily gradual escalation of the dose will be conducted with the oral suspension. Eight subjects will participate in each cohort. Four ascending dose levels are planned. Within each cohort 6 subjects will be randomised to receive AZD5718 and 2 subjects randomised to receive placebo. Each subject will receive one dose of AZD5718 or placebo on the first dosing day (Day 1, single ascending dose, SAD) and on Days 3 to 10 (multiple ascending dose, MAD). On Day 2 no dose will be given to the subject. In total each subject will receive 9 doses. Dosing for each ascending dose cohort will proceed after the SRC has evaluated the safety, tolerability and other relevant data of a completed cohort. The subjects will stay at the study site until 48 hours post-dose and will return 7 to 10 days after dosing for a follow-up visit. Each subject will be involved in the study for 7 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated, written informed consent prior to any study specific procedures
2. Healthy male Japanese subjects aged 18-50 years with suitable veins for cannulation or repeated venipuncture. A subject will be considered as Japanese if:

   * both of his parents and all grandparents are Japanese,
   * he was born in Japan and have a Japanese passport, and
   * he has not lived outside Japan for more than 10 years.
3. Have a body mass index (BMI) between 18 and 30 kg/m2 inclusive and weigh at least 50 kg and no more than 100 kg inclusive.
4. Provision of signed, written and dated informed consent for optional genetic/biomarker research. If a subject declines to participate in the genetic component of the study, there will be no penalty or loss of benefit to the subject. The subject will not be excluded from other aspects of the study described in this protocol.

Exclusion Criteria:

1. History of any clinically important disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
2. History or presence of gastrointestinal, hepatic or renal disease or any other condition known to interfere with absorption, distribution, metabolism or excretion of drugs.
3. Any clinically important illness, medical/surgical procedure or trauma within 4 weeks of the first administration of investigational medicinal product (IMP).
4. Any clinically important abnormalities in clinical chemistry, hematology or urinalysis results as judged by the Investigator.
5. Any positive result on Screening for serum hepatitis B surface antigen, hepatitis C antibody and human immunodeficiency virus (HIV).
6. Suspicion or known Gilbert's syndrome.
7. Abnormal vital signs, after 10 minutes supine rest, at screening and check-in, defined as any of the following (repeat evaluations may be done once if the values for a subject are outside the designated range at screening and on Day -1):

   Systolic blood pressure < 90 mmHg or > 140 mmHg Diastolic blood pressure < 50 mmHg or > 90 mmHg Heart rate < 45 or > 90 beats per minute (bpm)
8. Any clinically important abnormalities in rhythm, conduction or morphology of the resting ECG and any clinically important abnormalities at screening and check-in in the 12-Lead ECG as considered by the Investigator that may interfere with the interpretation of QTc interval changes, including abnormal ST-T-wave morphology, particularly in the protocol defined primary lead or left ventricular hypertrophy. If deemed necessary, an ECG may be repeated once for each ECG measurement.
9. Prolonged QTcF > 450 ms or shortened QTcF < 340 ms or family history of long QT syndrome at screening and check-in. If deemed necessary, an ECG may be repeated once for each ECG measurement.
10. PR(PQ) interval shortening < 120 ms (PR > 110 ms but < 120 ms is acceptable if there is no evidence of ventricular pre-excitation) at screening and check-in. If deemed necessary, an ECG may be repeated once for each ECG measurement.
11. PR (PQ) interval prolongation (> 240 ms) intermittent second (Wenckebach block while asleep is not exclusive) or third degree atrioventricular (AV) block, or AV dissociation at screening and check-in. If deemed necessary, an ECG may be repeated once for each ECG measurement.
12. Persistent or intermittent complete bundle branch block (BBB), incomplete bundle branch block (IBBB), or intraventricular conduction delay (IVCD) with QRS > 110 ms. Subjects with QRS > 110 ms but < 115 ms are acceptable if there is no evidence of e.g., ventricular hypertrophy or pre-excitation, at screening and check-in. If deemed necessary, an ECG may be repeated once for each ECG measurement.
13. Known or suspected history of drug abuse as judged by the Investigator.
14. Current smokers or those who have smoked or used nicotine products (including e-cigarettes within the previous 3 months).
15. History of alcohol abuse or excessive intake of alcohol as judged by the Investigator.
16. Positive screen for drugs of abuse or cotinine (nicotine) at screening and check-in (excluding cotinine).
17. History of severe allergy/hypersensitivity or ongoing clinically important allergy/hypersensitivity, as judged by the Investigator or history of hypersensitivity to drugs with a similar chemical structure or class to AZD5718.
18. Excessive intake of caffeine-containing drinks or food (e.g., coffee, tea, chocolate,) as judged by the Investigator.
19. Use of drugs with enzyme inducing properties such as St John's Wort within 3 weeks prior to the first administration of IMP.
20. Use of any prescribed or non-prescribed medication including antacids, analgesics (other than paracetamol/acetaminophen), herbal remedies, megadose vitamins (intake of 20 to 600 times the recommended daily dose) and minerals during the 2 weeks prior to the first administration of investigational product or longer if the medication has a long half-life.
21. Plasma donation within 1 month of Screening or any blood donation/blood loss > 500 mL during the 3 months prior to Screening.
22. Has received another new chemical entity (defined as a compound which has not been approved for marketing in the US) within 30 days or at least 5 half-lives (whichever is longer) of the first administration of investigational drug in this study. Note: subjects consented and screened, but not randomized in this study or a previous phase I study, are not excluded.
23. Subjects who have previously received AZD5718.
24. Involvement of any Astra Zeneca, PAREXEL or study site employee or their close relatives.
25. Judgment by the Investigator that the subject should not participate in the study if they have any ongoing or recent (i.e., during the Screening period) minor medical complaints that may interfere with the interpretation of study data or are considered unlikely to comply with study procedures, restrictions and requirements.
26. Subjects who are vegans or have medical dietary restrictions.
27. Subjects who cannot communicate reliably with the study team.
28. Vulnerable subjects, e.g., kept in detention, protected adults under guardianship, trusteeship, or committed to an institution by governmental or juridical order.

    In addition, any of the following is regarded as a criterion for exclusion from the genetic research:
29. Previous bone marrow transplant.
30. Non-leukocyte depleted whole blood transfusion within 120 days of the date of the genetic sample collection.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2018-01-16 (Actual); Primary Completion 2018-06-12 (Actual); Study Completion 2018-06-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with Adverse Events (AEs) due to AZD5817 | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the adverse events as a variable of safety and tolerability of AZD5718 following oral administration of single and multiple ascending doses. Adverse Events will be collected from the start of randomization throughout the treatment period up to and including the follow-up visit. Serious adverse events (SAEs) will be recorded from the time of informed consent.
Supine vital sign (Systolic Blood pressure [BP]) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the vital sign as a variable of safety and tolerability variable of AZD5718 following oral administration of single and multiple ascending doses.
Supine vital sign (pulse rate) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the vital sign as a variable of safety and tolerability of AZD5718 following oral administration of single and multiple ascending doses.
Number of participants with abnormal findings in electrocardiograms (ECGs) (safety ECGs, digital ECGs [dECG]) | From baseline up to follow-up (7 to 10 days post-(final) dose). For dECG: Days 1 to 12
  To assess any clinically important abnormalities in the cardiovascular system functioning as a variable of safety and tolerability of AZD5718 following oral administration of single and multiple ascending doses. A 12-lead 10-second safety ECG will be performed with the Schiller Cardiovit CS-200 recorder immediately following all scheduled dECGs. 12-lead continuous dECG will be recorded over at least 5 minutes with the Schiller Cardiovit CS-200 recorder and transmitted to the AstraZeneca central dECG repository, according to AstraZeneca ECG Center´s standard procedures for settings, recording, and transmission of dECGs. For dECG, QTcF (QT interval corrected for heart rate using Fridericia's formula) will be calculated as QTcF =(QT*(RR/1000)^(-1/3)), where RR (the time between corresponding points on 2 consecutive R waves on ECG) is presented in milliseconds. Heart rate (HR) will also be calculated, based on the RR interval.
Number of participants with abnormal cardiac telemetry | From baseline up to Day 10
  To assess any clinically important abnormalities in the cardiovascular system functioning (heart beat/rythm) using 2-lead real-time telemetry ECG as a variable of safety and tolerability of AZD5718 following oral administration of single and multiple ascending doses. The telemetry monitoring system will be reviewed by the Investigator or research nurse and paper printouts of any clinically important events will be stored as source data.
Number of participants with abnormal findings in physical examinations | From baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess any clinically important abnormal findings in physical conditions as a variable of safety and tolerability of AZD5718 following oral administration of single and multiple ascending doses. The complete physical examinations include an assessment of the general appearance, skin, cardiovascular, respiratory, abdomen, head, and neck (including ears, eyes, nose, and throat), lymph nodes, thyroid, musculoskeletal and neurological systems. The brief physical examinations include an assessment of the general appearance, skin, cardiovascular system, respiratory and abdomen. Any new or aggravated clinically relevant abnormal medical finding at a physical examination as compared with the baseline assessment will be reported as an adverse event.
Laboratory assessment: Hematology (leukocyte count) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the leukocyte count as a variable of safety and tolerability of AZD5718 following oral administration of single and multiple ascending doses.
Supine vital sign (diastolic BP) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the vital sign as a variable of safety and tolerability of AZD5718 following oral administration of single and multiple ascending doses.
Laboratory assessment: Clinical chemistry (sodium) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the clinical chemistry value (sodium) as a variable of safety and tolerability of AZD5718, following oral administration of single and multiple ascending doses.
Laboratory assessment: Urinalysis (glucose) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess urinalysis (glucose) as a variable of safety and tolerability of AZD5718, following oral administration of single and multiple ascending doses.
Laboratory assessment: Hematology (Red blood cell [RBC] count) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the RBC count as a variable of safety and tolerability of AZD5718 following oral administration of single and multiple ascending doses.
Laboratory assessment: Hematology (Hemoglobin [Hb]) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the Hb as a criterion of safety and tolerability variable of AZD5718 following oral administration of single and multiple ascending doses.
Laboratory assessment: Hematology (Hematocrit [HCT]) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the HCT as a variable of safety and tolerability of AZD5718 following oral administration of single and multiple ascending doses.
Laboratory assessment: Hematology (Mean corpuscular volume [MCV]) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the MCV as a variable of safety and tolerability of AZD5718 following oral administration of single and multiple ascending doses.
Laboratory assessment: Hematology (Mean corpuscular hemoglobin [MCH]) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the MCH as a variable of safety and tolerability of AZD5718 following oral administration of single and multiple ascending doses.
Laboratory assessment: Hematology (Mean corpuscular hemoglobin concentration [MCHC]) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the MCHC as a variable of safety and tolerability variable of AZD5718 following oral administration of single and multiple ascending doses.
Laboratory assessment: Clinical chemistry (potassium) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the clinical chemistry value (potassium) as a variable of safety and tolerability of AZD5718, following oral administration of single and multiple ascending doses.
Laboratory assessment: Clinical chemistry (urea) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the clinical chemistry value (urea) as a variable of safety and tolerability of AZD5718, following oral administration of single and multiple ascending doses.
Laboratory assessment: Clinical chemistry (creatinine) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the clinical chemistry value (creatinine) as a variable of safety and tolerability of AZD5718, following oral administration of single and multiple ascending doses.
Laboratory assessment: Clinical chemistry (albumin) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the clinical chemistry value (albumin) as a variable of safety and tolerability of AZD5718, following oral administration of single and multiple ascending doses.
Laboratory assessment: Clinical chemistry (calcium) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the clinical chemistry value (calcium) as a variable of safety and tolerability of AZD5718, following oral administration of single and multiple ascending doses.
Laboratory assessment: Clinical chemistry (phosphate) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the clinical chemistry value (phosphate) as a variable of safety and tolerability of AZD5718, following oral administration of single and multiple ascending doses.
Laboratory assessment: Clinical chemistry (glucose (fasting)) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the clinical chemistry value (glucose (fasting)) as a variable of safety and tolerability of AZD5718, following oral administration of single and multiple ascending doses.
Laboratory assessment: Clinical chemistry (insulin) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the clinical chemistry value (insulin) as a variable of safety and tolerability of AZD5718, following oral administration of single and multiple ascending doses.
Laboratory assessment: Clinical chemistry (fibrinogen) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the clinical chemistry value (fibrinogen) as a variable of safety and tolerability of AZD5718, following oral administration of single and multiple ascending doses.
Laboratory assessment: Clinical chemistry (thyroid-stimulating hormone) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the clinical chemistry value (thyroid-stimulating hormone) as a variable of safety and tolerability of AZD5718, following oral administration of single and multiple ascending doses.
Laboratory assessment: Urinalysis (blood) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess urinalysis (blood) as a variable of safety and tolerability of AZD5718, following oral administration of single and multiple ascending doses. If urinalysis is positive for blood, a microscopy test will be performed to assess RBC, white blood cell [WBC], casts [cellular, granular, hyaline]).
Laboratory assessment: Urinalysis (protein) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess urinalysis (protein) as a variable of safety and tolerability of AZD5718, following oral administration of single and multiple ascending doses. If urinalysis is positive for protein, a microscopy test will be performed to assess RBC, WBC, casts [cellular, granular, hyaline]).
Laboratory assessment: Urinalysis (urine creatinine) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess urinalysis (urine creatinine) as a variable of safety and tolerability of AZD5718, following oral administration of single and multiple ascending doses.
Laboratory assessment: Hematology (Differential Count) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the differential count as a variable of safety and tolerability of AZD5718 following oral administration of single and multiple ascending doses.
Laboratory assessment: Hematology (Platelets) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the platelets as a variable of safety and tolerability of AZD5718 following oral administration of single and multiple ascending doses.
Laboratory assessment: Hematology (Reticulocytes absolute count) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the reticulocytes absolute count as a variable of safety and tolerability of AZD5718 following oral administration of single and multiple ascending doses.
Laboratory assessment: Clinical chemistry (High sensitivity-C-reactive protein [CRP]) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the clinical chemistry value (CRP) as a variable of safety and tolerability of AZD5718, following oral administration of single and multiple ascending doses.
Laboratory assessment: Clinical chemistry (Free T4) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the clinical chemistry value (Free T4) as a variable of safety and tolerability of AZD5718, following oral administration of single and multiple ascending doses.
Laboratory assessment: Clinical chemistry (Alkaline phosphatase [ALP]) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the clinical chemistry value (ALP) as a variable of safety and tolerability of AZD5718, following oral administration of single and multiple ascending doses.
Laboratory assessment: Clinical chemistry (Alanine aminotransferase [ALT]) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the clinical chemistry value (ALT) as a variable of safety and tolerability of AZD5718, following oral administration of single and multiple ascending doses.
Laboratory assessment: Clinical chemistry (Aspartate aminotransferase [AST]) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the clinical chemistry value (AST) as a variable of safety and tolerability of AZD5718, following oral administration of single and multiple ascending doses.
Laboratory assessment: Clinical chemistry (Gamma glutamyl transpeptidase [GGT]) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the clinical chemistry value (GGT) as a variable of safety and tolerability of AZD5718, following oral administration of single and multiple ascending doses.
Laboratory assessment: Clinical chemistry (Total Bilirubin) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the clinical chemistry value (total bilirubin) as a variable of safety and tolerability of AZD5718, following oral administration of single and multiple ascending doses.
Laboratory assessment: Clinical chemistry (Unconjugated bilirubin) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the clinical chemistry value (unconjugated bilirubin) as a variable of safety and tolerability of AZD5718, following oral administration of single and multiple ascending doses.
Laboratory assessment: Clinical chemistry (Glutamate dehydrogenase) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the clinical chemistry value (glutamate dehydrogenase) as a variable of safety and tolerability of AZD5718, following oral administration of single and multiple ascending doses.
Laboratory assessment: Clinical chemistry (Lactate dehydrogenase [LDH]) | Change from baseline up to follow-up (7 to 10 days post-(final) dose)
  To assess the clinical chemistry value (LDH) as a variable of safety and tolerability of AZD5718, following oral administration of single and multiple ascending doses.

SECONDARY OUTCOMES:
Plasma PK assessment: Observed maximum plasma concentration (Cmax) assessment for AZD5817 after single and repeated oral dosing | Day 1 and Day 10: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 32 and 48 hours (Day 3 pre-dose) post-dose, Day 4-9 pre morning dose
  To assess Cmax of AZD5718 after single and repeated oral dosing.
Plasma PK assessment: Time to reach peak or maximum observed concentration following drug administration (tmax) assessment for AZD5817 after single and repeated oral dosing | Day 1 and Day 10: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 32 and 48 hours (Day 3 pre-dose) post-dose, Day 4-9 pre morning dose
  To assess tmax of AZD5718 after single and repeated oral dosing.
Plasma PK assessment: Terminal rate constant (λZ) assessment for AZD5817 after single and repeated oral dosing | Day 1 and Day 10: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 32 and 48 hours (Day 3 pre-dose) post-dose, Day 4-9 pre morning dose
  To assess λZ of AZD5718 after single and repeated oral dosing. λZ will be estimated by log-linear least-squares regression of the terminal part of the concentration-time curve.
Plasma PK assessment: Terminal half-life (t½λz) assessment for AZD5817 after single and repeated oral dosing | Day 1 and Day 10: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 32 and 48 hours (Day 3 pre-dose) post-dose, Day 4-9 pre morning dose
  To assess t½λz of AZD5718 after single and repeated oral dosing. t½λz will be estimated as (ln2)/λZ.
Plasma PK assessment: Area under the plasma concentration-time curve from time zero to 24 hours after dosing (AUC(0-24)) assessment for AZD5817 after single and repeated oral dosing | Day 1 and Day 10: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 32 and 48 hours (Day 3 pre-dose) post-dose, Day 4-9 pre morning dose
  To assess AUC(0-24) of AZD5718 after single and repeated oral dosing.
Plasma PK assessment: Area under the plasma concentration-curve from time zero to the time of last quantifiable analyte concentration (AUC(0-last)) assessment for AZD5817 after single and repeated oral dosing | Day 1 and Day 10: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 32 and 48 hours (Day 3 pre-dose) post-dose, Day 4-9 pre morning dose
  To assess AUC(0-last) of AZD5718 after single and repeated oral dosing.
Plasma PK assessment: Area under the plasma concentration-curve over the dosing interval (AUC(0-τ)) assessment for AZD5817 after single and repeated oral dosing | Day 1 and Day 10: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 32 and 48 hours (Day 3 pre-dose) post-dose, Day 4-9 pre morning dose
  To assess AUC(0-τ) of AZD5718 after single and repeated oral dosing.
Plasma PK assessment: Area under the concentration-time curve from time zero extrapolated to infinity (AUC) assessment for AZD5817 after single and repeated oral dosing | Day 1 and Day 10: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 32 and 48 hours (Day 3 pre-dose) post-dose, Day 4-9 pre morning dose
  To assess AUC of AZD5718 after single and repeated oral dosing. AUC is estimated by AUC(0-last) + Clast/λZ where Clast is the last observed quantifiable concentration.
Plasma PK assessment: Apparent total body clearance of drug from plasma after extravascular administration (CL/F) assessment for AZD5817 after single and repeated oral dosing | Day 1 and Day 10: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 32 and 48 hours (Day 3 pre-dose) post-dose, Day 4-9 pre morning dose
  To assess CL/F of AZD5718 after single and repeated oral dosing.
Plasma PK assessment: Mean Residence Time (MRT) assessment for AZD5817 after single and repeated oral dosing | Day 1 and Day 10: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 32 and 48 hours (Day 3 pre-dose) post-dose
  To assess MRT of AZD5718 after single and repeated oral dosing.
Plasma PK assessment: Apparent volume of distribution for parent drug at terminal phase (extravascular administration), (Vz/F) assessment for AZD5817 after single and repeated oral dosing | Day 1 and Day 10: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 32 and 48 hours (Day 3 pre-dose) post-dose, Day 4-9 pre morning dose
  To assess Vz/F of AZD5718 after single and repeated oral dosing. Vz/F will be estimated by dividing the apparent clearance (CL/F) by λZ.
Plasma PK assessment: Observed minimum concentration, (Cmin) assessment for AZD5817 after single and repeated oral dosing (Day 10) | Day 10: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 32 and 48 hours (Day 3 pre-dose) post-dose
  To assess Cmin of AZD5718 after single and repeated oral dosing. Cmin will be taken directly from the individual concentration-time curve.
Plasma PK assessment: Observed average concentration (Cavg) assessment for AZD5817 after single and repeated oral dosing (Day 10) | Day 10: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 32 and 48 hours (Day 3 pre-dose) post-dose
  To assess Cavg of AZD5718 after single and repeated oral dosing. Cavg will be taken directly from the individual concentration-time curve.
Plasma PK assessment: Accumulation ratio (Rac Cmax) assessment for AZD5817 after single and repeated oral dosing | Day 1 and Day 10: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 32 and 48 hours (Day 3 pre-dose) post-dose
  To assess Rac Cmax of AZD5718 after single and repeated oral dosing. Rac Cmax will be calculated as Cmax Day 10/ Cmax Day 1.
Plasma PK assessment: Accumulation ratio (Rac AUC) assessment for AZD5817 after single and repeated oral dosing | Day 1 and Day 10: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 32 and 48 hours (Day 3 pre-dose) post-dose
  To assess Rac AUC of AZD5718 after single and repeated oral dosing. Rac AUC will be calculated as AUCτ Day 10/ AUCτ Day 1.
Plasma PK assessment: Temporal change parameter in systemic exposure (TCP) assessment for AZD5817 after single and repeated oral dosing | Day 1 and Day 10: pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 12, 16, 24, 32 and 48 hours (Day 3 pre-dose) post-dose, Day 4-9 pre morning dose
  To assess TCP of AZD5718 after single and repeated oral dosing. TCP will be calculated as AUCτDay 10/AUCDay 1.
Urine PK assessment: Cumulative amount of unchanged drug excreted in urine from time zero to the last sampling interval (Ae(0-last)) assessment for AZD5817 after single and repeated oral dosing | Day 10 pooled 0-3, 3-6, 6-9, 9-12 hours and 12-24 hours urine
  To assess Ae(0-last) of AZD5718 after single and repeated oral dosing.
Urine PK assessment: Fraction of dose excreted unchanged into the urine from time zero to the last sampling interval measured time point for an analyte (Fe(0-last)) assessment for AZD5817 after single and repeated oral dosing | Day 10 pooled 0-3, 3-6, 6-9, 9-12 hours and 12-24 hours urine
  To assess Fe(0-last) of AZD5718 after single and repeated oral dosing. Fe(0-last) will be estimated by dividing Ae(0-last) by dose.
Urine PK assessment: Renal clearance of drug from plasma (CLR) assessment for AZD5817 after single and repeated oral dosing | Day 10 pooled 0-3, 3-6, 6-9, 9-12 hours and 12-24 hours urine
  To assess CLR of AZD5718 after single and repeated oral dosing. CLR will be estimated by dividing Ae(0-last) by AUC(0-t)).
PD parameter: urine Leukotriene E4 (LTE4) assessment for AZD5817 after single and repeated oral dosing | Day -1 (spot sample), Day 1 and Day 10 spot sample pre-dose and pooled 0-3, 3-6, 6-9 and 9-12 hours urine, spot sample at 24, 36 hours post-dose, Day 3-9: spot sample pre-dose
  To evaluate the PD of AZD5718, by assessment of urine LTE4 (u-LTE4), after single and repeated oral dosing.

CONTACTS AND LOCATIONS:
Overall Officials: David Han, Dr, Principal Investigator — PAREXEL Early Phase Clinical Unit-Los Angeles
Locations (1):
- Research Site, Glendale, California, United States